CLINICAL TRIAL: NCT05493124
Title: Clinical Study of Manpixiao in the Treatment of Chronic Atrophic Gastritis
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Dr. Xia Ding, Professor, Beijing University of Chinese Medicine
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-ZXFZJJ-035
Record Dates: First submitted 2022-07-29; First posted 2022-08-09 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2021-09

CONDITIONS: Chronic Atrophic Gastritis
MeSH Terms: conditions — Gastritis, Atrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manpixiao treatment group (Experimental): A traditional Chinese medicine composition (has applied for Chinese patent)，Take 17.15g daily, twice in the morning and evening, for a total of 24 weeks
  Interventions: Drug: Manpixiao
- Blank treatment group (No Intervention)
- Active comparator (Active Comparator): Including treated with Chinese patent drugs such as Weifuchun and morodan, or treated with antacids, motivational drugs, gastric mucosal protectants, vitamins, folic acid, selenium containing preparations and other drugs. Take it according to the instructions.
  Interventions: Drug: Active comparator

INTERVENTIONS:
Drug: Manpixiao — A traditional Chinese medicine composition
  Arms: Manpixiao treatment group
Drug: Active comparator — Other drugs that may have therapeutic effects
  Arms: Active comparator

SUMMARY:
To explore the efficacy and safety of "Manpixiao" in the treatment of Chronic Atrophic Gastritis.

ELIGIBILITY:
Inclusion Criteria:

* The age is 18-75 years old, regardless of gender;
* Before treatment, the patients were diagnosed as chronic atrophic gastritis (with intestinal metaplasia and dysplasia) by gastroscopy and pathological examination, which met the criteria of the Chinese consensus on chronic gastritis (2017, Shanghai);
* Sign the informed consent form.

Exclusion Criteria:

* Patients with autoimmune gastritis (chronic atrophic gastritis type A), peptic ulcer (a1-h2), reflux esophagitis, gastric polyps, hypertrophic gastritis and other diseases;
* Patients with high-grade intraepithelial neoplasia of gastric mucosa, suspected malignant change of gastrointestinal mucosal lesions, and gastrointestinal tumors;
* Patients with malignant tumors who have undergone surgery, radiotherapy and chemotherapy in recent 5 years;
* Patients with primary diseases such as heart, brain, lung, hematopoietic system and malignant tumors, and subjects with severe diabetes;
* Patients with chronic liver and kidney dysfunction before treatment, including ALT > 1.5 times the upper limit of normal value, blood creatinine (CR) > 1.5 times the upper limit of normal value, and platelets lower than 1.5 times the lower limit of normal value;
* Disabled subjects specified by law (blind, deaf, dumb, intellectual, mental, physical disabilities);
* The description of self symptoms is unclear or the investigation is not the author;
* Have a history of alcohol abuse;
* Allergic constitution or a history of allergy to multiple drugs (more than two or known ingredients in the drug);
* Pregnant or lactating women;
* According to the judgment of the researcher, other reasons should not be selected.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological improvement rate of gastric mucosa | The enrollment inspection shall be completed within one month before enrollment; The examination after treatment should be carried out within 1 month after the completion of treatment.
  Pathological diagnosis of gastric mucosal tissue samples obtained by gastroscopy

SECONDARY OUTCOMES:
Gastric mucosal status under gastroscope | The enrollment inspection shall be completed within one month before enrollment; The examination after treatment should be carried out within 1 month after the completion of treatment.
  For the color of gastric mucosa, spots, erosion, bleeding, reduced folds, visible blood vessels and mucosal texture, 0, 1, 2 and 3 points are given according to the levels of none, I, II and III respectively, and 0 and 1 points are given according to the presence or absence of bile reflux. According to the gastroscopy report, score the patients' microscopic results before and after treatment, and take the result change as the secondary index of curative effect. A lower score means a better result.
Score of main symptoms of stomach system | They were evaluated on the day of enrollment and the day of the end of the treatment process
  Adopt the "table of main symptoms of stomach system based on doctor's report", the specific contents are: epigastric (epigastric) pain, epigastric (epigastric) distension, epigastric (epigastric) blockage, heartburn, acid reflux, belching, anorexia, reduced appetite. Score 0, 1, 2 and 3 points for the severity of each single symptom (none, mild, moderate and severe). The total score of symptoms is the sum of the individual scores. By comparing the changes of individual symptom scores and total symptom scores between groups, lower scores mean better results.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Dongfang Hospital, Beijing University of Chinese Medicine, Beijing
  - Dongzhimen Hospital, Beijing University of TCM, Beijing
  - Zaozhuang Hospital, Beijing University of Chinese Medicine, Beijing

IPD SHARING:
Plan to Share IPD: Yes
Obtained by asking the first or correspondent author if necessary
Supporting Information: CSR
Time Frame: One year after the completion of the study
Access Criteria: Obtained by asking the first or correspondent author if necessary

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/24/NCT05493124/Prot_SAP_ICF_000.pdf